CLINICAL TRIAL: NCT04165850
Title: Open Label Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of Ciprofloxacin/Celecoxib Combination in Patients With ALS
Brief Title: Open Label Study to Evaluate Ciprofloxacin/Celecoxib Combination in Patients With ALS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeuroSense Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NST002
Record Dates: First submitted 2019-11-13; First posted 2019-11-18 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2019-11

CONDITIONS: Amyotrophic Lateral Sclerosis; ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Celecoxib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fixed dose Ciprofloxacin and Celecoxib (Experimental): Fixed dose Ciprofloxacin and Celecoxib capsule to be taken thrice daily, total dose 909mg/day
  Interventions: Drug: Fixed dose combination Ciprofloxacin/Celecoxib

INTERVENTIONS:
Drug: Fixed dose combination Ciprofloxacin/Celecoxib — Fixed dose Ciprofloxacin and Celecoxib capsule to be taken thrice daily, total dose 909mg/day
  Other Names: PrimeC

SUMMARY:
This is an open label, off label study, to provide interested ALS patients with Ciprofloxacin/Celecoxib fixed dose combination, while assessing safety and tolerability and routine disease progression measures (ALSFRS-R and Vital Capacity).

DETAILED DESCRIPTION:
Patients will be prescribed a fixed dose combination of Ciprofloxacin and Celecoxib to be taken thrice daily, and will be monitored for safety and tolerability. Additionally, routine disease progression measures will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and willing to sign an Informed Consent Form (ICF)
2. Males or females between the ages of 18 and 75 years of age, inclusive
3. Diagnosis of familial or sporadic ALS (defined as meeting the laboratory-supported probable, probable, or definite criteria for a diagnosis of ALS according to the World Federation of Neurology El Escorial criteria)
4. Disease duration after first symptom less than 3 years prior to baseline
5. Patients may be treated in parallel with Riluzole and/or Edaravone; 30 days of stable use prior to enrollment is required
6. Upright forced vital capacity (FVC) ≥ 50% of predicted for age, height, weight and sex at screening
7. Patient is able to swallow tablets/ capsules
8. A caregiver (if one is needed)
9. Female patients must be post-menopausal (≥ 1 year) OR sterilized, OR if of childbearing potential (i.e., females who have had their first period unless they are anatomically or physiologically incapable to become pregnant), must have a negative pregnancy test, and agree to use contraceptive drugs or devices (e.g., diaphragm plus spermicide, or oral contraceptives) for the duration of the study and 10 weeks after the last treatment dose AND require male partners to use a condom during sexual intercourse

Exclusion Criteria:

1. A past history of adverse reaction/hypersensitivity to either NSAIDs, celecoxib or fluoroquinolones, ciprofloxacin
2. Any known clinically significant abnormal gastric mucosal erosion, ulcer or tumor or/and GI disorder
3. Known history of clinically significant impairment of renal function (creatinine ≥ 1.5)
4. Known or suspected congestive heart and/or coronary heart disease, previous history of myocardial infarction, uncontrolled arterial hypertension, or rhythm abnormalities requiring permanent treatment
5. Known history of QT/QTc prolongation, Torsade de pointes (TdP) (e.g. heart failure, hypokalemia, family history of Long QT syndrome) and the use of concomitant medications that prolong the QT/QTc interval
6. Known or suspected diagnosis or family history of epilepsy
7. Presence at screening of any medically significant cardiac, pulmonary, musculoskeletal, or psychiatric illness that might interfere with the patient's ability to comply with study procedures or that might confound the interpretation of clinical safety data, including, but not limited to:

   1. Mean systolic blood pressure >180 mm Hg; mean diastolic blood pressure >100 mm Hg (measurements taken after few min rest) that persist on 3 successive measurements taken at least 2 minutes apart
   2. NYHA Class II or greater congestive heart failure
   3. Chronic obstructive pulmonary disease or asthma requiring daily use of bronchodilator medications
   4. Poorly controlled or brittle diabetes mellitus
   5. Cognitive impairment, related to ALS or otherwise, sufficient to impair patient's ability to understand and/or comply with study procedures and provide informed consent
8. Patient who is treated with chronic aspirin or NSAIDs, and is at risk if stopped. Clopidogrel is allowed and can replace Aspirin.
9. Female who is pregnant or breastfeeding or with intention of becoming pregnant during the course of the study
10. Any impairment or social circumstance that, in the opinion of the Investigator, would render the patient not suitable to participate in the study
11. Patient, patient's parent(s), or patient's legal guardian(s) is/are unable to understand the nature, scope, and possible consequences of the study
12. Patient is participating in (or plans to participate in) any other investigational drug trial, or plans to be exposed to any other investigational agent, device and/or procedure, from 30 days prior to Screening through study completion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-01-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with one or more treatment-emergent adverse events | 15 months
  Treatment emergent adverse event is any medical event associated with the drug
Number of patients who discontinued treatment prematurely | 15 months
  Number of patients whose treatment is stopped prematurely for any reason
Number of patients who discontinued treatment prematurely due to adverse events | 15 months
  Number of patients whose treatment is stopped prematurely specifically due to adverse events
Number of patients with significant abnormal laboratory values | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Drory, MD, Principal Investigator — Sourasky Medical Center
Locations (1):
- Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No